CLINICAL TRIAL: NCT06953817
Title: The Effect of Kangaroo Care Education Given to Pregnant Women in the Third Trimester on Mother-Infant Bonding, Maternal and Neonatal Comfort: A Randomized Controlled Trial
Brief Title: The Effect of Kangaroo Care Education on Mother-Infant Bonding, Maternal and Neonatal Comfort
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Emel AVÇİN, Lecturer Dr, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Emel Avcin Kangaroo Care
Record Dates: First submitted 2025-04-15; First posted 2025-05-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Kangaroo Care; Pregnant; Bonding; Comfort
Keywords: Kangaroo care; Neonatal; Mother-Infant Bonding; Neonatal Comfort

STUDY DESIGN:
Intervention Model Description: Randomized controlled and quasi-experimental research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo care group (Experimental): In the initial visit, kangaroo care education will be provided to the pregnant women through a guide/presentation prepared by the researchers, accompanied by hands-on training with a baby. Later, the pregnant women will practice it with a non-real baby. The kangaroo care video prepared by the researchers will be sent to the pregnant women. A chart will be provided to track how many times the pregnant women watch the video. Throughout the study, messages regarding kangaroo care will be sent to the mothers. After being informed by the mothers/fathers that labor has started, they will be visited at the hospital within the first 24 hours. The infant information form, mother-infant bonding scale, kangaroo care comfort scale, and neonatal comfort behavior scale will be completed. Pregnant women will be asked to continue kangaroo care for four weeks after delivery, and at the end of this period, data collection forms will be completed via WhatsApp.
  Interventions: Behavioral: Kangaroo Care Intervention Group
- Control group (No Intervention): No intervention will be applied to the control group. The pregnant women will be informed about their expected delivery date and will be instructed to notify the researchers when labor begins. After being informed by the mothers/fathers that labor has started, they will be visited within the first 24 hours at the hospital, and the infant information form, mother-infant bonding scale, kangaroo care comfort scale, and neonatal comfort behavior scale will be completed. Four weeks later, the data collection forms will be sent via WhatsApp, and the participants will be asked to complete them. At the end of the study, it will be announced that the study has concluded. At the conclusion of the study, the mothers in this group will also receive a guide and video about the importance and application of kangaroo care via WhatsApp.

INTERVENTIONS:
Behavioral: Kangaroo Care Intervention Group — The mother should wear a comfortable outfit that can be easily opened at the front, and attention should be given to the mother's privacy. The infant should be covered with a light blanket. While applying kangaroo care, the baby may be completely naked, or the baby may wear items such as a hat, diaper, and socks. The kangaroo care position involves placing the baby upright between the mother's breasts. The newborn's abdomen should be positioned at the level of the mother's epigastric region. While performing kangaroo care, the mother should ensure that the baby's face is visible and that the baby's head is not in extreme extension or excessive flexion. During the procedure, care should be taken to ensure that the baby can breathe comfortably while on the mother's chest. The pregnant women will be instructed to practice kangaroo care intermittently for 30 minutes.
  Arms: Kangaroo care group

SUMMARY:
Kangaroo care encompasses early and continuous skin-to-skin contact, frequent and regular breastfeeding, early discharge from the hospital, and other supportive care practices necessary for the infant . Through kangaroo care, the transition of newborns from intrauterine to extrauterine life is facilitated, and a strong and secure bond between the mother and the newborn is established. Kangaroo care, which does not require any additional equipment or special preparation, is a safe method that can be easily and frequently implemented due to its numerous benefits. Since maternal and neonatal health affects not only the family but also public health, maternal and neonatal comfort is considered to be of great importance. Kangaroo care is believed to contribute positively to the enhancement of this comfort and the strengthening of the mother-infant bond. Despite the well-documented benefits of kangaroo care in the literature, its implementation in our country has not reached the desired level. This study is planned to determine the effect of kangaroo care education provided to pregnant women in the third trimester on mother-infant bonding and maternal and neonatal comfort.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Pregnant Women:

* Aged 18 years or older,
* Primiparous (first pregnancy),
* Between 35-38 weeks of gestation,
* Able to speak Turkish and/or without communication barriers,
* At least a primary school graduate,
* A healthy pregnancy,
* Good health status during and after delivery,
* No contraindications for providing kangaroo care,
* No physical and/or mental health issues,
* No infectious diseases transmitted through contact,
* Willing to participate in the study,
* Use of WhatsApp application,
* Pregnant women expecting a single baby will be included in the study.

Inclusion Criteria for the Infant:

* Full-term,
* No need for oxygen support,
* No congenital anomalies,
* No infectious diseases,
* Stable general condition.

Exclusion Criteria:

* Exclusion Criteria for Pregnant Women:
* Multiparity,
* Foreign nationals, migrants, or those with communication difficulties,
* High-risk pregnancies,
* Physical and/or mental health issues,
* Presence of an infectious disease transmitted through contact,
* Refusal to participate in the study,
* Non-users of phone and/or WhatsApp application,
* Pregnant women expecting multiple babies will be excluded from the study.

Exclusion Criteria during Data Collection:

* Women who no longer wish to continue in the study after volunteering,
* Women who cannot be reached via WhatsApp and/or phone,
* Women whose infants experience death (exitus),
* Women whose infants have conditions preventing the application of kangaroo care will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since it will be conducted with pregnant women in the third trimester
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Mother-Infant Bonding in Pregnant Women Who Received Kangaroo Care Education in the Third Trimester | At the time of first participation in the study in the third trimester, within the first 24 hours after delivery, and 4 weeks after delivery
  After being informed by the mother/father that labor has started, they will be visited at the hospital within the first 24 hours. During this visit, it will be inquired whether the mother has applied kangaroo care, and she will be encouraged to do so. The infant information form, mother-infant bonding scale will be completed. As the final follow-up, a video call will be conducted with the mother 4 weeks later, and she will be asked to complete the survey forms sent via WhatsApp.
Evaluation of Maternal Comfort in Pregnant Women Who Received Kangaroo Care Education in the Third Trimester | At the time of first participation in the study in the third trimester, within the first 24 hours after delivery, and 4 weeks after delivery
  The infant information form, mother kangaroo care comfort scale will be completed. As the final follow-up, a video call will be conducted with the mother 4 weeks later, and she will be asked to complete the survey forms sent via WhatsApp.
Evaluation of Neonatal Comfort in Pregnant Women Who Received Kangaroo Care Education in the Third Trimester | Newborn comfort behaviors will be evaluated within the first 24 hours after birth and again at 4 weeks postpartum.
  The infant information form, neonatal comfort behaviour scale will be completed. As the final follow-up, a video call will be conducted with the mother 4 weeks later, and she will be asked to complete the survey forms sent via WhatsApp.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL AVÇİN, Doctor, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)